CLINICAL TRIAL: NCT01910220
Title: Study to Assess the Safety and Bioeffect of REGN1033 (SAR391786)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Regeneron Pharmaceuticals (Industry)
Collaborators: Sanofi (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: R1033-HV-1223
Record Dates: First submitted 2013-07-25; First posted 2013-07-29 (Estimated); Last update posted 2014-11-10 (Estimated); Status verified 2014-11

CONDITIONS: Healthy Volunteers

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (4):
- Group 1 (Placebo Comparator): placebo
  Interventions: Other: placebo
- Group 2 (Experimental): REGN1033 (SAR391786)
  Interventions: Drug: REGN1033 (SAR391786)
- Group 3 (Placebo Comparator): placebo + exercise regimen
  Interventions: Other: placebo
- Group 4 (Experimental): REGN1033 (SAR391786) + exercise regimen
  Interventions: Drug: REGN1033 (SAR391786)

INTERVENTIONS:
Drug: REGN1033 (SAR391786)
  Arms: Group 2; Group 4
Other: placebo
  Arms: Group 1; Group 3

SUMMARY:
This is a study to assess the safety and bioeffect of REGN1033 (SAR391786) in healthy volunteers.

ELIGIBILITY:
Inclusion Criteria:

1. Males and postmenopausal females aged 60 years and older with no significant health issues or clinically significant abnormal laboratory values.
2. Low activity lifestyle
3. Diet and exercise adherence

Exclusion Criteria:

1. Significant concomitant illness such as, but not limited to cardiac, renal, rheumatologic, gastrointestinal, hematological, skeletal/muscular, neurologic, psychiatric, endocrine, metabolic or immunological disease.
2. Participation in any clinical trial within 6 months prior to screening.
3. Hospitalization, immobilization, or major surgical procedure requiring general anesthesia within 6 months prior to screening, or any planned surgical procedures during the study period.
4. Limb amputation (except for toes) and/or any fracture within 6 months.

The above information is not intended to contain all considerations relevant to a patient's potential participation in a clinical trial and not all inclusion/ exclusion criteria are listed.

Min Age: 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 125 (Actual)
Dates: Start 2013-08; Primary Completion 2014-06 (Actual); Study Completion 2014-10 (Actual)

PRIMARY OUTCOMES:
Percent change in total lean mass | At week 12
  The primary endpoint is percent change in total lean mass at week 12 (day 85)

SECONDARY OUTCOMES:
Number of TEAEs | day 1 to day 141
  Number of treatment-emergent adverse events (TEAEs) from day 1 (baseline) to day 141 (end of study)
Appendicular lean mass by DXA | At week 12
  Appendicular lean mass by DXA (dual energy X-ray absorptiometry) at week 12

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trial Management, Study Director — Regeneron Pharmaceuticals
Locations (5):
- United States (5):
  - Gainesville, Florida
  - Orlando, Florida
  - Boston, Massachusetts
  - St Louis, Missouri
  - Athens, Ohio